CLINICAL TRIAL: NCT03057106
Title: A Randomized Trial of Durvalumab and Tremelimumab ± Platinum-Based Chemotherapy in Patients With Metastatic (Stage IV) Squamous or Non-Squamous Non-Small Cell Lung Cancer (NSCLC)
Brief Title: Durvalumab and Tremelimumab ± Platinum-Based Chemotherapy in Patients With Metastatic Squamous or Non-Squamous NSCLC
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Canadian Cancer Trials Group (Network)
Collaborators: AstraZeneca (Industry); Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other); National Health and Medical Research Council, Australia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BR34
Record Dates: First submitted 2017-02-15; First posted 2017-02-17 (Actual); Results first posted 2022-02-09 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Lung Cancer Metastatic
MeSH Terms: interventions — durvalumab; tremelimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Durvalumab and Tremelimumab (Active Comparator): Durvalumab q4 weeks until PD + Tremelimumab q 4 wk x 4 doses
  Interventions: Drug: Durvalumab; Drug: Tremelimumab
- Platinum based chemotherapy + Durvalumab + Tremelimumab (Active Comparator): 4 cycles platinum plus gem or pem + Durva + Treme (q 3 wk x 4 cycles)
  Followed by:
  Squamous Cell: Maintenance Durva q 4 wk until PD Non-Squamous Cell: Pemetrexed + Durva q 4 wk until PD
  Interventions: Drug: Durvalumab; Drug: Tremelimumab; Drug: Platinum-Based Drug

INTERVENTIONS:
Drug: Durvalumab — MEDI4736
Drug: Tremelimumab — Tremelimumab
Drug: Platinum-Based Drug — Pemetrexed, cisplatin, carboplatin or gemcitibine
  Arms: Platinum based chemotherapy + Durvalumab + Tremelimumab

SUMMARY:
Durvalumab is a new type of drug for many kinds of cancer. It is considered "immunotherapy" and not "chemotherapy". Laboratory tests show that it works by allowing the immune system to detect cancer and reactivate the immune response. This may help to slow down the growth of cancer or may cause cancer cells to die. Durvalumab has been shown to shrink tumours in animals and has been studied in more than 5000 people and seems promising.

Tremelimumab is a new type of drug for various types of cancers. It works in a similar way to durvalumab and may improve the effect of durvalumab. Tremelimumab may also help slow the growth of the cancer cells or may cause cancer cells to die. It has been shown to shrink tumours in animals and has been studied in over 1200 people and seems promising.

DETAILED DESCRIPTION:
Combinations of durvalumab and tremelimumab have also been studied. While the combination has been studied in over 200 people, it is not clear if it can offer better results when it is combined with chemotherapy.

Recently, immunotherapies that target the PD-1/PD-L1 axis have shown promise in treating patients with non-small cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically and/or cytologically confirmed diagnosis of squamous or non-squamous, non-small cell carcinoma of the lung. Patients with poorly differentiated tumours will only be eligible if NSCLC is confirmed by immunohistochemistry markers (TTF1/P63 or P40/CK5). Patients with known sensitizing EGFR mutations or known ALK-fusion are not eligible.
* Patients must have stage IV disease according to the 8th TNM version staging.
* Patients must have an adequate histopathology specimen and must consent to release this specimen for protocol required testing. This is a mandatory component of the study.
* Patient must consent to provision of samples of blood in order that the specific correlative marker assays proscribed may be conducted.
* All patients must have measurable disease as defined by RECIST 1.1 All radiology studies must be performed within 28 days prior to randomization (within 35 days if negative).

The criteria for defining measurable disease are as follows:

* CT scan (with slice thickness of 5 mm) ≥ 10 mm --> longest diameter
* Physical exam (using calipers) ≥ 10 mm
* Lymph nodes by CT scan ≥ 15 mm --> measured in short axis

Measurable lesions must be outside a previous radiotherapy field if they are the sole site of disease, unless disease progression has been documented.

* Patients must be 18 years of age or older.
* ECOG performance status of 0 or 1.
* Absolute neutrophils ≥ 1.5 x 10^9/L
* Platelets ≥ 100 x 10^9/L
* Hemoglobin ≥ 90 g/L
* Bilirubin ≤ 1.5 x UNL (upper limit of normal)
* AST and ALT ≤ 2.5 x UNL (if liver metastases are present, ≤5 x UNL) Creatinine < 1.25 UNL or Creatinine clearance ≥ 45 mL/min
* Cytotoxic Chemotherapy: Patients may not have received prior cytotoxic chemotherapy for advanced/metastatic disease.
* Adjuvant Chemotherapy: Patients may have had prior adjuvant therapy for completely resected disease, providing it has been completed at least 12 months prior to randomization.
* Patients treated with concurrent chemotherapy/radiation regimens for unresectable locally advanced Stage III disease will be eligible providing it has been completed at least 12 months prior to randomization.
* Other Systemic Therapy: Patients may not have received prior EGFR or alk inhibitors. Patients may not have received prior treatment with immune-based therapy, including durvalumab and tremelimumab vaccines or oncolytic viral therapy. Patients must have recovered from any reversible treatment related toxicities prior to randomization.
* Prior external beam radiation is permitted provided a minimum of 14 days (2 weeks) have elapsed between the last dose of radiation and date of randomization. Concurrent radiotherapy is not permitted.

Patients must have recovered from any acute toxic effects from radiation prior to randomization.

* Patients must have recovered from any acute toxic effects from radiation prior to randomization.
* Surgery: Previous surgery is permitted provided that wound healing has occurred and at least 14 days have elapsed (major surgery) prior to randomization.
* Patient must be able (i.e. sufficiently fluent) and willing to complete the quality of life and health economics questionnaires.
* Patient consent must be appropriately obtained in accordance with applicable local and regulatory requirements.
* Patients must be accessible for treatment and follow-up. All randomized patients must be followed and treated at participating centres.
* In accordance with CCTG policy, protocol treatment is to begin within 2 working days of patient randomization.
* Female patients of childbearing potential who are sexually active with a non-sterilized male partner must use at least one highly effective method of contraception while on study and for 6 months after the last dose of durvalumab and tremelimumab or for 3 months after the last dose of durvalumab alone

Exclusion Criteria:

* Patients with a history of other malignancies, except: adequately treated non-melanoma skin cancer, curatively treated in-situ cancer of the cervix, or other solid tumours curatively treated with no evidence of disease for ≥ 3 years. Patients with a history of other malignancies detected at an early stage and whom the investigator believes have been curatively treated and are at low risk of recurrence MAY be eligible. Contact CCTG to discuss eligibility prior to enrolling.
* Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease (e.g. colitis or Crohn's disease), diverticulitis with the exception of diverticulosis, celiac disease or other serious gastrointestinal chronic conditions associated with diarrhea), systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome (granulomatosis with polyangiitis), rheumatoid arthritis, hypophysitis, uveitis, etc., within the past 3 years prior to the start of treatment. The following are exceptions to this criterion:

  * Patients with alopecia.
  * Patients with Grave's disease, vitiligo or psoriasis not requiring systemic treatment (within the last 2 years).
  * Patients with hypothyroidism (e.g. following Hashimoto syndrome) stable on hormone replacement.
* History of primary immunodeficiency, history of allogenic organ transplant that requires therapeutic immunosuppression and the use of immunosuppressive agents within 28 days of randomization* or a prior history of severe (grade 3 or 4) immune mediated toxicity from other immune therapy or grade ≥ 3 infusion reaction.
* Live attenuated vaccination administered within 30 days prior to randomization
* History of hypersensitivity to durvalumab or tremelimumab or any excipient. Patients who have received other treatment or other antibodies must not have had intolerable toxicity or required steroids to manage toxicity.
* Mean QT interval corrected for heart rate using Fridericia's formula (QTcF) ≥ 470 msec in screening ECG measured using standard institutional method or history of familial long QT syndrome.
* Patients who have untreated and/or uncontrolled cardiovascular conditions and/or have symptomatic cardiac dysfunction (unstable angina, congestive heart failure, myocardial infarction within the previous year or cardiac ventricular arrhythmias requiring medication, history of 2nd or 3rd degree atrioventricular conduction defects). Patients with a significant cardiac history, even if now controlled, should have a LVEF ≥ 45%. (Note: patients with uncomplicated controlled hypertension do not require LVEF measurement in the absence of other significant cardiac history)
* Concurrent treatment with other investigational drugs or anti-cancer therapy
* Patients with untreated brain or meningeal metastases are not eligible. Patients with treated CNS disease who have radiologic AND clinical evidence of stable brain metastases, with no evidence of cavitation or hemorrhage in the brain lesion, are eligible providing that they are asymptomatic and do not require corticosteroids (must have discontinued steroids at least 1 week prior to randomization).
* Pregnant or Lactating Women: Women of childbearing potential must have a pregnancy test (urine or serum) proven negative within 14 days prior to randomization. If urine test is positive, pregnancy testing may then include an ultrasound to rule-out pregnancy if a false-positive is suspected. For example, when beta-human chorionic gonadotropin is high and partner is vasectomized, it may be associated with tumour production of hCG, as seen with some cancers. Patient will be considered eligible if an ultrasound is negative for pregnancy. Men and women of child-bearing potential must agree to use adequate contraception.
* Patients with serious illnesses or medical conditions which would not permit the patient to be managed according to the protocol (including corticosteroid administration), or would put the patient at risk. This includes but is not limited to:

  * Contraindications to the use of pemetrexed, gemcitabine, cisplatin and/or carboplatin (consult product monograph);
  * History of significant neurologic or psychiatric disorder which would impair the ability to obtain consent or limit compliance with study requirements;
  * Active infection requiring systemic therapy; (including any patient known to have active hepatitis B, hepatitis C or human immunodeficiency virus (HIV) or tuberculosis);
  * Active peptic ulcer disease or gastritis;
  * Known pneumonitis or pulmonary fibrosis with clinically significant impairment of pulmonary function.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 301 (Actual)
Dates: Start 2017-03-28 (Actual); Primary Completion 2020-02-24 (Actual); Study Completion 2025-12-30 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Natasha Leighl, Study Chair — Princess Margaret Hospital, Toronto, ON Canada
Locations (49):
- Australia (19):
  - Campbelltown Hospital, Campbelltown, New South Wales
  - Coffs Habour Health Campus - NCCI, Coffs Harbour, New South Wales
  - Concord Repatriation General Hospital, Concord, New South Wales
  - Nepean Hospital, Kingswood, New South Wales
  - St. George Hospital, Cancer Care Centre, Kogarah, New South Wales
  - The Tweed Hospital, Lismore, New South Wales
  - Liverpool Cancer Therapy Centre, Liverpool Hospital, Liverpool, New South Wales
  - Prince of Wales Hospital, Randwick, New South Wales
  - Princess Alexandra Hospital, Brisbane, Queensland
  - The Prince Charles Hospital, Chermside, Queensland
  - Mater Research Institute South Brisbane, South Brisbane, Queensland
  - Gold Coast University Hospital, Southport, Queensland
  - Toowoomba Hospital, Toowoomba, Queensland
  - Royal Hobart Hospital, Hobart, Tasmania
  - Ballarat Health Services, Ballarat, Victoria
  - Epworth HealthCare - Richmond, Richmond, Victoria
  - Border Medical Oncology, Wodonga, Victoria
  - Saint John of God Hospital Subiaco, Subiaco, Western Australia
  - St. Vincent's Hospital, Victoria Park
- Canada (30):
  - Cross Cancer Institute, Edmonton, Alberta
  - BCCA - Fraser Valley Cancer Centre, Surrey, British Columbia
  - BCCA - Vancouver Cancer Centre, Vancouver, British Columbia
  - Horizon Health Network, Fredericton, New Brunswick
  - The Moncton Hospital, Moncton, New Brunswick
  - The Vitalite Health Network - Dr. Leon Richard, Moncton, New Brunswick
  - Regional Health Authority B, Zone 2, Saint John, New Brunswick
  - Cambridge Memorial Hospital, Cambridge, Ontario
  - Health Sciences North, Greater Sudbury, Ontario
  - Juravinski Cancer Centre at Hamilton Health Sciences, Hamilton, Ontario
  - Kingston Health Sciences Centre, Kingston, Ontario
  - Grand River Regional Cancer Centre, Kitchener, Ontario
  - Stronach Regional Health Centre at Southlake, Newmarket, Ontario
  - Ottawa Hospital Research Institute, Ottawa, Ontario
  - Algoma District Cancer Program, Sault Ste. Marie, Ontario
  - Niagara Health System, St. Catharines, Ontario
  - North York General Hospital, Toronto, Ontario
  - Humber River Regional Hospital, Toronto, Ontario
  - Michael Garron Hospital, Toronto, Ontario
  - University Health Network, Toronto, Ontario
  - Windsor Regional Cancer Centre, Windsor, Ontario
  - PEI Cancer Treatment Centre, Charlottetown, Prince Edward Island
  - Hopital de la Cite-de-la-Sante, Laval, Quebec
  - CHUM-Centre Hospitalier de l'Universite de Montreal, Montreal, Quebec
  - The Jewish General Hospital, Montreal, Quebec
  - CHU de Quebec-Hopital l'Enfant-Jesus (HEJ), Québec, Quebec
  - University Institute of Cardiology and, Québec, Quebec
  - Centre hospitalier universitaire de Sherbrooke, Sherbrooke, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Leighl NB, Laurie SA, Goss GD, Hughes BGM, Stockler M, Tsao MS, Hwang DM, Joubert P, Kulkarni S, Blais N, Joy AA, Mates M, Rana P, Yadav SK, Underhill C, Lee C, Bradbury PA, Hiltz A, Dancey J, Ding K, Vera-Badillo F; Canadian Cancer Trials Group Lung Disease Site and the Australasian Lung Cancer Trials Group. CCTG BR34: A Randomized Phase 2 Trial of Durvalumab and Tremelimumab With or Without Platinum-Based Chemotherapy in Patients With Metastatic NSCLC. J Thorac Oncol. 2022 Mar;17(3):434-445. doi: 10.1016/j.jtho.2021.10.023. Epub 2021 Nov 17. PMID 34800700

RESULTS

PARTICIPANT FLOW:
Groups:
- Platinum Based Chemotherapy + Durvalumab + Tremelimumab: 4 cycles platinum plus gem or pem + Durva + Treme (q 3 wk x 4 cycles)
  Followed by:
  Squamous Cell: Maintenance Durva q 4 wk until PD Non-Squamous Cell: Pemetrexed + Durva q 4 wk until PD
  Durvalumab: MEDI4736
  Tremelimumab: Tremelimumab
  Platinum-Based Drug: Pemetrexed, cisplatin, carboplatin or gemcitibine
Period: Overall Study
Arm/Group | Durvalumab and Tremelimumab | Platinum Based Chemotherapy + Durvalumab + Tremelimumab
Started (4 patient refused study treatment) | 149 (1 patient refused the treatment) | 148 (3 patients refused the treatment)
Completed | 149 | 148
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: ITT population, included 4 patients who refused the study treatments.
Groups:
- Total: Total of all reporting groups
Arm/Group | Durvalumab and Tremelimumab | Platinum Based Chemotherapy + Durvalumab + Tremelimumab | Total
Number analyzed (Participants) | 150 | 151 | 301
Age, Categorical [Count of Participants; unit: Participants]
  Age: <=18 years | 0 | 0 | 0
  Age: Between 18 and 65 years | 86 | 69 | 155
  Age: >=65 years | 64 | 82 | 146
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 69 | 70 | 139
  Male | 81 | 81 | 162
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 2
  Asian | 6 | 7 | 13
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 4 | 0 | 4
  White | 138 | 138 | 276
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 3 | 5
Smoking history [Count of Participants; unit: Participants]
  Never smoke | 14 | 12 | 26
  Ever smoked | 136 | 139 | 275
Histology type [Count of Participants; unit: Participants]
  Non-squamous | 123 | 123 | 246
  Squamous | 27 | 28 | 55
ECOG Performance Status [Count of Participants; unit: Participants] — 0: Fully active, able to carry on all pre-disease performance without restriction.
  1: Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work.
  Participants
    0 | 45 | 47 | 92
    1 | 105 | 104 | 209

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: time from randomization to the date of death
Time Frame: 33 months
Population: ITT population, included patients who refused the study treatments (4 patients)
Measure: Median (90% Confidence Interval); unit: Months
Arm/Group | Durvalumab and Tremelimumab | Platinum Based Chemotherapy + Durvalumab + Tremelimumab
Number analyzed (Participants) | 150 | 151
Months | 14.1 [10.6 to 18.3] | 16.6 [12.6 to 19.1]
Statistical Analysis 1: Comparison: Durvalumab and Tremelimumab vs Platinum Based Chemotherapy + Durvalumab + Tremelimumab; Test type: Superiority; p = 0.46, Log Rank — 2-sided, adjusted for stratification factors at rtandomization; Hazard Ratio (HR) = 0.88, 90% CI 2-sided [0.67 to 1.16]

2. Secondary Outcome: Progression-free Survival Using RECIST 1.1
Description: time from randomization to the date of the first documented disease progression. Progression was defined as: at least a 20% increase in the sum of diameters of measured lesions taking as references the smallest sum of diameters recorded on study (including baseline) AND an absolute increase of ≥5 mm, or appearance of new lesions.
Time Frame: 33 months
Population: ITT population, included the 4 patents who refused study treatments.
Measure: Median (90% Confidence Interval); unit: Months
Arm/Group | Durvalumab and Tremelimumab | Platinum Based Chemotherapy + Durvalumab + Tremelimumab
Number analyzed (Participants) | 150 | 151
Months | 3.22 [2.73 to 5.13] | 7.72 [5.52 to 8.54]
Statistical Analysis 1: Comparison: Durvalumab and Tremelimumab vs Platinum Based Chemotherapy + Durvalumab + Tremelimumab; Test type: Superiority; p = 0.0035, Log Rank — 2-sided, adjusted for stratification factors at randomization; Adjusted for stratification factors at randomization; Hazard Ratio (HR) = 0.67, 95% CI 2-sided [0.52 to 0.88]

3. Secondary Outcome: Objective Response Rate Using RECIST 1.1 and iRECIST
Description: proportion of patients with a documented complete response, partial response (CR + PR) based on iRECIST criteria. The primary estimate of ORR will be based on all patients randomized, and compared using Cochran- Mantel-Haeszel test stratified by stratification factors at randomization between the study new treatment and the standard control arms.
Time Frame: 33 months
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | Durvalumab and Tremelimumab | Platinum Based Chemotherapy + Durvalumab + Tremelimumab
Number analyzed (Participants) | 150 | 151
Participants
  Partial Response | 44 | 64
  Stable Disease | 47 | 53
  Progressive Disease | 53 | 25
  Inevaluable | 6 | 9
Statistical Analysis 1: Comparison: Durvalumab and Tremelimumab vs Platinum Based Chemotherapy + Durvalumab + Tremelimumab; Test type: Superiority; p = 0.033, Cochran-Mantel-Haenszel — 2-sided, adjusted for stratification factors at randomization; Odds Ratio (OR) = 1.69, 95% CI 2-sided [1.04 to 2.76]

ADVERSE EVENTS:
Time Frame: 33 months
Description: Adverse events graded according to CTCAE Version 4.0.
Arm/Group | Durvalumab and Tremelimumab | Platinum Based Chemotherapy + Durvalumab + Tremelimumab
All-Cause Mortality (participants affected / at risk) | 80/149 | 77/148
Serious Adverse Events (participants affected / at risk) | 84/149 | 102/148
Other Adverse Events (participants affected / at risk) | 149/149 | 148/148
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Durvalumab and Tremelimumab (N=149) | Platinum Based Chemotherapy + Durvalumab + Tremelimumab (N=148)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 12 (12)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 7 (7)
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 1 (1)
Asystole (Cardiac disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 4 (4)
Atrial flutter (Cardiac disorders) | 2 (2) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1) | 1 (1)
Chest pain - cardiac (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 3 (3) | 2 (2)
Pericardial tamponade (Cardiac disorders) | 2 (2) | 0 (0)
Pericarditis (Cardiac disorders) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 2 (2)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 3 (3) | 3 (3)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 0 (0) | 2 (2)
Scleral disorder (Eye disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 2 (2)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 14 (14) | 11 (11)
Constipation (Gastrointestinal disorders) | 2 (2) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 16 (16) | 10 (10)
Duodenal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Enterocolitis (Gastrointestinal disorders) | 4 (4) | 2 (2)
Gastric hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 2 (2) | 1 (1)
Nausea (Gastrointestinal disorders) | 4 (4) | 5 (5)
Oral hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Other gastrointestinal disorders (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 2 (2) | 2 (2)
Vomiting (Gastrointestinal disorders) | 4 (4) | 4 (4)
Death NOS (General disorders) | 0 (0) | 2 (2)
Fatigue (General disorders) | 1 (1) | 2 (2)
Fever (General disorders) | 5 (5) | 11 (11)
Flu like symptoms (General disorders) | 1 (1) | 2 (2)
Infusion related reaction (General disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1)
Other general disorders, administration site conditions (General disorders) | 1 (1) | 1 (1)
Pain (General disorders) | 1 (1) | 1 (1)
Sudden death NOS (General disorders) | 1 (1) | 0 (0)
Allergic reaction (Immune system disorders) | 0 (0) | 2 (2)
Autoimmune disorder (Immune system disorders) | 0 (0) | 1 (1)
Cytokine release syndrome (Immune system disorders) | 0 (0) | 1 (1)
Other immune system disorders (Immune system disorders) | 2 (2) | 6 (6)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1)
Gallbladder infection (Infections and infestations) | 0 (0) | 1 (1)
Joint infection (Infections and infestations) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 11 (11) | 12 (12)
Other infections and infestations (Infections and infestations) | 0 (0) | 6 (6)
Sepsis (Infections and infestations) | 2 (2) | 2 (2)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 0 (0) | 3 (3)
Upper respiratory infection (Infections and infestations) | 3 (3) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Alanine aminotransferase increased (Investigations) | 4 (4) | 4 (4)
Alkaline phosphatase increased (Investigations) | 3 (3) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 4 (4) | 6 (6)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1)
Creatinine increased (Investigations) | 1 (1) | 4 (4)
GGT increased (Investigations) | 3 (3) | 1 (1)
Lipase increased (Investigations) | 4 (4) | 4 (4)
Neutrophil count decreased (Investigations) | 0 (0) | 4 (4)
Platelet count decreased (Investigations) | 0 (0) | 10 (10)
Serum amylase increased (Investigations) | 2 (2) | 2 (2)
Weight loss (Investigations) | 0 (0) | 1 (1)
White blood cell decreased (Investigations) | 0 (0) | 2 (2)
Acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 4 (4)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Myositis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Other neoplasms benign, malignant and unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 13 (13) | 18 (18)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Dysesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Edema cerebral (Nervous system disorders) | 1 (1) | 1 (1)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Facial nerve disorder (Nervous system disorders) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 1 (1)
Intracranial hemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Lethargy (Nervous system disorders) | 1 (1) | 0 (0)
Other nervous system disorders (Nervous system disorders) | 0 (0) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Radiculitis (Nervous system disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 3 (3) | 1 (1)
Stroke (Nervous system disorders) | 4 (4) | 1 (1)
Transient ischemic attacks (Nervous system disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Confusion (Psychiatric disorders) | 2 (2) | 0 (0)
Delirium (Psychiatric disorders) | 2 (2) | 2 (2)
Acute kidney injury (Renal and urinary disorders) | 2 (2) | 3 (3)
Other renal and urinary disorders (Renal and urinary disorders) | 0 (0) | 1 (1)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Chylothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 4 (4)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Other respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 2 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 7 (7)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Other skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 5 (5) | 7 (7)
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 2 (2)
Other vascular disorders (Vascular disorders) | 0 (0) | 1 (1)
Superficial thrombophlebitis (Vascular disorders) | 0 (0) | 1 (1)
Superior vena cava syndrome (Vascular disorders) | 0 (0) | 1 (1)
Thromboembolic event (Vascular disorders) | 7 (7) | 9 (9)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Durvalumab and Tremelimumab (N=149) | Platinum Based Chemotherapy + Durvalumab + Tremelimumab (N=148)
Sinus tachycardia (Cardiac disorders) | 2 (2) | 8 (8)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 8 (8)
Tinnitus (Ear and labyrinth disorders) | 6 (6) | 17 (17)
Hypothyroidism (Endocrine disorders) | 19 (19) | 18 (18)
Blurred vision (Eye disorders) | 10 (10) | 10 (10)
Other eye disorders (Eye disorders) | 5 (5) | 15 (15)
Watering eyes (Eye disorders) | 1 (1) | 20 (20)
Abdominal pain (Gastrointestinal disorders) | 26 (26) | 29 (29)
Bloating (Gastrointestinal disorders) | 4 (4) | 11 (11)
Colitis (Gastrointestinal disorders) | 11 (11) | 8 (8)
Constipation (Gastrointestinal disorders) | 60 (60) | 84 (84)
Diarrhea (Gastrointestinal disorders) | 50 (50) | 72 (72)
Dry mouth (Gastrointestinal disorders) | 15 (15) | 19 (19)
Dyspepsia (Gastrointestinal disorders) | 8 (8) | 18 (18)
Dysphagia (Gastrointestinal disorders) | 4 (4) | 9 (9)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 13 (13) | 14 (14)
Mucositis oral (Gastrointestinal disorders) | 12 (12) | 22 (22)
Nausea (Gastrointestinal disorders) | 60 (60) | 101 (101)
Vomiting (Gastrointestinal disorders) | 36 (36) | 54 (54)
Chills (General disorders) | 8 (8) | 11 (11)
Edema limbs (General disorders) | 21 (21) | 42 (42)
Fatigue (General disorders) | 105 (105) | 125 (125)
Fever (General disorders) | 22 (22) | 28 (28)
Flu like symptoms (General disorders) | 11 (11) | 17 (17)
Non-cardiac chest pain (General disorders) | 31 (31) | 24 (24)
Pain (General disorders) | 24 (24) | 30 (30)
Other immune system disorders (Immune system disorders) | 5 (5) | 11 (11)
Lung infection (Infections and infestations) | 12 (12) | 15 (15)
Other infections and infestations (Infections and infestations) | 12 (12) | 7 (7)
Skin infection (Infections and infestations) | 2 (2) | 8 (8)
Upper respiratory infection (Infections and infestations) | 27 (27) | 18 (18)
Urinary tract infection (Infections and infestations) | 6 (6) | 16 (16)
Bruising (Injury, poisoning and procedural complications) | 2 (2) | 10 (10)
Creatinine increased (Investigations) | 1 (1) | 8 (8)
Weight gain (Investigations) | 3 (3) | 12 (12)
Weight loss (Investigations) | 41 (41) | 37 (37)
Anorexia (Metabolism and nutrition disorders) | 68 (68) | 78 (78)
Dehydration (Metabolism and nutrition disorders) | 4 (4) | 12 (12)
Hypokalemia (Metabolism and nutrition disorders) | 15 (15) | 17 (17)
Hypomagnesemia (Metabolism and nutrition disorders) | 5 (5) | 17 (17)
Hyponatremia (Metabolism and nutrition disorders) | 9 (9) | 6 (6)
Arthralgia (Musculoskeletal and connective tissue disorders) | 25 (25) | 22 (22)
Back pain (Musculoskeletal and connective tissue disorders) | 57 (57) | 55 (55)
Bone pain (Musculoskeletal and connective tissue disorders) | 18 (18) | 17 (17)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 16 (16) | 16 (16)
Flank pain (Musculoskeletal and connective tissue disorders) | 6 (6) | 9 (9)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 9 (9) | 17 (17)
Myalgia (Musculoskeletal and connective tissue disorders) | 9 (9) | 10 (10)
Neck pain (Musculoskeletal and connective tissue disorders) | 12 (12) | 12 (12)
Other musculoskeletal and connective tissue disorder (Musculoskeletal and connective tissue disorders) | 8 (8) | 8 (8)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 33 (33) | 41 (41)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 11 (11) | 7 (7)
Dizziness (Nervous system disorders) | 16 (16) | 32 (32)
Dysgeusia (Nervous system disorders) | 13 (13) | 23 (23)
Headache (Nervous system disorders) | 29 (29) | 41 (41)
Paresthesia (Nervous system disorders) | 9 (9) | 8 (8)
Peripheral sensory neuropathy (Nervous system disorders) | 13 (13) | 30 (30)
Anxiety (Psychiatric disorders) | 26 (26) | 24 (24)
Confusion (Psychiatric disorders) | 4 (4) | 9 (9)
Depression (Psychiatric disorders) | 16 (16) | 15 (15)
Insomnia (Psychiatric disorders) | 46 (46) | 56 (56)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 15 (15)
Cough (Respiratory, thoracic and mediastinal disorders) | 65 (65) | 79 (79)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 93 (93) | 95 (95)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 11 (11)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 8 (8)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 9 (9)
Other respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 11 (11) | 12 (12)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 19 (19) | 24 (24)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 8 (8)
Alopecia (Skin and subcutaneous tissue disorders) | 8 (8) | 23 (23)
Dry skin (Skin and subcutaneous tissue disorders) | 10 (10) | 15 (15)
Other skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 10 (10) | 20 (20)
Pruritus (Skin and subcutaneous tissue disorders) | 39 (39) | 44 (44)
Rash acneiform (Skin and subcutaneous tissue disorders) | 8 (8) | 15 (15)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 42 (42) | 45 (45)
Hypertension (Vascular disorders) | 9 (9) | 15 (15)
Hypotension (Vascular disorders) | 7 (7) | 13 (13)
Thromboembolic event (Vascular disorders) | 12 (12) | 14 (14)

LIMITATIONS AND CAVEATS:
The small sample size may prevent the study to find identify the biomarker defined subgroup that may be benefit from the study treatment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-02-19): https://cdn.clinicaltrials.gov/large-docs/06/NCT03057106/Prot_000.pdf
  • Statistical Analysis Plan (2019-11-01): https://cdn.clinicaltrials.gov/large-docs/06/NCT03057106/SAP_001.pdf